CLINICAL TRIAL: NCT04182919
Title: "Efficacy and Safety of Phlai Capsule Compared to Placebo as the Treatment in Allergic Rhinitis Patients"
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Collaborators: Government Pharmaceutical Organization (Unknown)
Responsible Party: Principal Investigator, Minh Phuoc Hoang, MD, Principal Investigator, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COA-CREC036/2019
Record Dates: First submitted 2019-11-26; First posted 2019-12-02 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Allergic Rhinitis
Keywords: Zingiber cassumunar; Phlai; compound D; herbal medicine; allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: Participant in each arm will take medication provided by care providers who also do not know what kind of this medication
Who Masked: Participant, Care Provider
Masking Description: Participant, care provider and investigator, outcomes assessor in each site do not know what kind of medication in each package.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Phlai 2 capsules (compound D 8 mg) od evening after meal x 4 weeks
  Interventions: Drug: Phlai
- Arm 2 (Experimental): Phlai 1 capsules (compound D 4 mg) and placebo 1 capsule od evening after meal x 4 weeks
  Interventions: Drug: Phlai; Drug: Placebo oral capsule
- Arm 3 (Placebo Comparator): Placebo 2 capsules od evening after meal x 4 weeks
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Phlai — Each capsule contains 4 mg compound D. Using orally in the evening everyday in 4 weeks
  Other Names: Zingiber cassumunar
  Arms: Arm 1; Arm 2
Drug: Placebo oral capsule — Like Phlai capsule extract : :PVP K30, Calcium carbonate, Dibasic calcium phosphate, Sodium starch glycolate, Colloidal silicon dioxide, Ethanol 96%, Purified water, Magnesium stearate. Not having compound D. Using orally in the evening everyday in 4 weeks
  Arms: Arm 2; Arm 3

SUMMARY:
Background: Zingiber cassumunar Roxb., frequently known as Phlai in Thai, has been safely used as an antihistaminic and anti-inflammatory drug in Thai traditional medicine. Individual with allergic rhinitis may have positive response to Phlai.

Objective: Investigators assessed the efficacy and safety of Phlai as a treatment for allergic rhinitis Design: The study was a 1-month, double-blind, randomized, parallel-group, intent-to-treat, multicenter, controlled trial in 267 patients at 7 hospitals in Thailand. Skin prick test-positive adults with allergic rhinitis ages 18 to 50 who were randomized into 3 groups (Phlai 8mg/d, Phlai 4mg/d, placebo).

Main outcome measures: Primary outcome was defined: improvement of total 5 symptoms scores (nasal obstruction, rhinorrhea, sneezing, itchy nose, itchy eyes) over a 4-week interval among Phlai 8mg/d, Phlai 4mg/d and placebo. Secondary endpoints were: assessments of rhinoconjunctivitis quality of life questionnaire, peak inspiratory nasal flow, nasal examination, adverse events, AST, ALT, Creatinine and BUN over a period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years old
* Allergic rhinitis following diagnostic criteria of ARIA guideline
* Reflective total 5 symptoms score 2-10 per day for 3 consecutive days (total score=15) and not greater than 10 in any days during the past week
* Positive skin prick test to at least one aeroallergen: wheal size ≥ 3 mm greater than negative control
* Not receiving intranasal corticosteroid + intra antihistamine for 2 weeks , intranasal corticosteroid for 2 weeks, systemic corticosteroid for 4 weeks, antihistamine for 1 week, nasal decongestant for 1 week and leukotriene receptor antagonists for 1 week

Exclusion Criteria:

* Serious medical underlying diseases e.g. COPD, Heart disease, Chronic renal failure, chronic hepatic failure
* Allergic rhinitis and asthma which require immunotherapy
* Receiving antidepressants, sedative, anxiolytic, opioids, neuroleptic
* Uncontrolled asthma which requires steroid inhaler, LABA and does not use leukotriene receptor antagonists
* Previous nasal surgery for nasal polyp, nasal septum deviation
* Acute or chronic rhinosinusitis
* Pregnancy and lactation (Urine pregnancy test is allowed and paid by researchers)
* Allergic to any kinds of herb
* Refusal to participation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 267 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Total five symptoms score (T5SS) | 24 hours
  T5SS: (nasal obstruction, rhinorrhea, sneezing, itchy nose, itchy eyes). For each symptom:
  0: no symptoms
  1. mild
  2. moderate
  3. severe. Participants assess T5SS everyday. Self assessment twice a day Bedtime : reflective symptoms score Morning :instantaneous symptoms score. The mean score of two assessment is the T5SS. Investigator will calculate the mean T5SS in the follow up

SECONDARY OUTCOMES:
Rhinoconjunctivitis Quality of Life Questionaire (RCQ-36) Thai version | 4 weeks
  This questionnaire is designed to find out how your health and well-being have been affected by rhinoconjunctivitis.
Peak inspiratory nasal flow (PNIF) | 2 weeks
  Use to measure nasal airflow during maximal inspiration
Nasal examination | 2 weeks
  Outcome assessor in each site will check the three symptoms: nasal swelling, pale and nasal discharge by anterior rhinoscopy
Adverse events | 2 weeks
  Sedation, dizziness, dry mouth, headache
AST Level | 4 weeks
  Liver function test
ALT Level | 4 weeks
  Liver function test
Creatinine level | 4 weeks
  Renal function test
BUN | 4 weeks
  Renal function test
Eosinophils blood level | 4 weeks
  CBC test
Lymphocyte blood level | 4 weeks
  CBC test
Hemoglobin | 4 weeks
  CBC test
Platelet level | 4 weeks
  CBC test

CONTACTS AND LOCATIONS:
Locations (1):
- Minh Phuoc Hoang, MD, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Will plan to share information when finishing study
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Plan to complete study in 2 years and will share the data after get publication